CLINICAL TRIAL: NCT07318909
Title: A Clinical Exploration Study of Adeno-Associated Virus Vector Expressing Human Phenylalanine Hydroxylase Gene in Adult Classical Phenylketonuria
Brief Title: To Evaluate the Safety and Efficacy of GS1168 Injection in Adult Phenylketonuria
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gritgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS1168-201
Record Dates: First submitted 2025-12-01; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group Arm of GS1168 (Experimental): Dose level 1, level 2 and level 3 will be administered
  Interventions: Drug: GS1168 injection

INTERVENTIONS:
Drug: GS1168 injection — The dose levels are as follows:
  1. A single intravenous administration of GS1168 injection at dose level 1;
  2. A single intravenous administration of GS1168 injection at dose level 2;
  3. A single intravenous administration of GS1168 injection at dose level 3.

SUMMARY:
This study is a single-arm, open-label, dose-escalation, exploratory study to evaluate the safety, tolerability, and efficacy of a single administration of GS1168 Injection in Chinese adult phenylketonuria (PKU) with PAH mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the purpose and risks of the study and voluntarily sign Informed Consent Forms (ICF).
2. Male or female, aged 18-55 years.
3. Diagnosis of PKU due to PAH mutation, and be inadequately controlled with current therapy (e.g., dietary management) in the judgement of the investigator.
4. Intolerant of unresponsive to available treatment such as Kuvan or Palynziq, and have come off the medication for at least 28 days prior to signing the ICF.
5. Ability and willingness to maintain dietary protein intake consistent with baseline
6. Male and female subjects of childbearing potential must agree to use effective contraception methods from signing ICF until at least 52 weeks after GS1168 infusion. Female subjects must not be breastfeeding.
7. Agree to avoid alcohol consumption from 30 days prior to GS1168 infusion until at least 52 weeks after infusion.
8. Ability to communicate well with the Investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Diagnosis of PKU due to other gene mutations.
2. Body weight ≥100 kg or Body Mass Index (BMI) ≥30 kg/m² at screening.
3. Presence of anti-AAV8 neutralizing antibody.
4. Abnormal liver function tests at screening:

   * ALT or AST >1.25 × Upper Limit of Normal (ULN)
   * GGT >1.25 × ULN
   * Total Bilirubin >1.5 × ULN
5. Abnormal laboratory findings at screening:

   * Hemoglobin <9 g/dL
   * Neutrophil count <1.0 × 10⁹/L
   * Platelet count <100 × 10⁹/L
   * Serum Creatinine ≥1.5 mg/dL (133 μmol/L)
   * Glycated Hemoglobin (HbA1c) >6% or Fasting Blood Glucose >6.1 mmol/L
6. Active or occult hepatitis B virus (HBV) infection, active hepatitis C virus (HCV) infection, positive Human Immunodeficiency Virus (HIV) antibodies and positive syphilis test.
7. Any severe conditions of respiratory, cardiovascular, gastrointestinal, renal, neurological, endocrine, immunological, hematological, psychiatric, etc.
8. History of malignancy.
9. Any other condition that, in the opinion of the Investigator, may affect subject compliance or render the subject unsuitable for participation in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event (AE), including serious adverse event (SAE) and adverse event of special interest (AESI) | Week 52
  Incidence of adverse event (AE), including serious adverse event (SAE) and adverse event of special interest (AESI) as assessed by CTCAE V5.0, from baseline to week 52

SECONDARY OUTCOMES:
Plasma Phe levels | Week 52
  Change from baseline in plasma level of Phe following GS1168 injection administration
Total protein intake | Week 52
  Change from baseline in total protein intake following GS1168 injection administration
Phenylketonuria Quality of Life (PKU-QOL) scores | Week 52
  Change in Phenylketonuria Quality of Life Questionnaire (PKU-QOL, Score range: 0-100, higher scores indicate worse outcomes.)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No